CLINICAL TRIAL: NCT01844011
Title: Promoting Fetal Movement Monitoring: Improving Birth Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Medical Center (Other)
Collaborators: First Candle Foundation (Unknown)
Responsible Party: Principal Investigator, Michael Mullen, Administration, Mercy Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MMC 2011-56
Record Dates: First submitted 2013-04-26; First posted 2013-05-01 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Fetal Kick Counting
Keywords: fetal movement; pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily electronic reminders (Experimental): Women in the intervention arm will be sent either daily text messages on the weekdays on their cell phone or emails on the weekdays reminding them to track kick counts on the chart.
  Interventions: Other: Daily electronic reminders
- Education only (No Intervention): All women enrolled in the trial will receive a paper-based kick count chart, will be educated in the use of the kick count chart, and will be instructed to keep track of their fetal movements on a daily basis.

INTERVENTIONS:
Other: Daily electronic reminders — Women in the intervention arm will be sent either daily text messages on the weekdays on their cell phone or emails on the weekdays reminding them to track kick counts on the chart
  Arms: Daily electronic reminders

SUMMARY:
The purpose of the study is to find out the best way to help pregnant women keep track of their baby's movements. During pregnancy, feeling your baby's movements is normal. A decrease in movement can indicate potential problems with your baby's well-being. This study will see if daily electronic reminders and kick count charts help women to better track their baby's movements over the last weeks of pregnancy.

DETAILED DESCRIPTION:
Pregnant women coming to the Hoffman and Associates or the Center for Advanced Fetal Care at Mercy Medical Center for their prenatal care and delivery may join this study. You must be able to receive daily text messages on your cell phone or have access to a computer to check daily emails in order to take part in the study. It is expected that 80 pregnant women will take part in this study. The study will end within a month after the delivery of your baby.

There is some evidence in the published literature suggesting that maternal monitoring of fetal movement may improve fetal mortality rates and infant health. Kick counting is a specific strategy to monitor fetal movement. Kick counts are typically performed in a daily 10-minute increment or until a specified number of "kicks" has been counted. In general, keeping track of kick counts begins in the 28th week of pregnancy, or earlier for high-risk pregnancies. Keeping track of kick counts allows the mother to monitor her baby's normal activity pattern and to identify when the baby's movement may decrease.

This study will be conducted to examine whether daily electronic reminders, sent using either cell phone text messages or computer-based emails, delivered in conjunction with the use of a paper-based kick count chart, increases the likelihood of completion of the paper-based kick count chart as well as knowledge regarding use of kick count methods compared to the paper-based kick count chart alone.

ELIGIBILITY:
Inclusion Criteria:

* 24-28 weeks pregnant
* able to receive daily text messages or emails
* 18 years of age or older
* willing to sign informed consent

Exclusion Criteria:

-unable to sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Completion of Paper Chart | 36 weeks pregnant-1 month status post delivery
  Completion of kick count charts at follow-up prenatal visits
Knowledge of kick counting post delivery | 36 weeks pregnant-1 month status post delivery
  Baseline questionnaire, including knowledge questions regarding monitoring baby's movement and kick count methods can be compared to post-education kick count knowledge questionnaire, week 36 questionnaire and end of study questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kathy J Helzlsouer, MD, Principal Investigator — Mercy Medical Center; Robert Atlas, MD, Principal Investigator — Mercy Medical Center
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States